CLINICAL TRIAL: NCT00192270
Title: A Prospective, Open-label, Phase II, Multi-center Study of the Safety, Tolerability and Immunogenicity of Influenza Virus Vaccine, Trivalent, Types A and B, Live Cold-adapted (CAIV-T) in Healthy Children, Aged 6 to 17 Years
Brief Title: Trial to Assess Safety, Tolerability, and Immunogenicity of Influenza Virus Vaccine, Trivalent, Types A and B, Live Cold-adapted (CAIV-T) in Healthy Children
Acronym: FluMist
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Raburn Mallory MD/ Sr Dir Clinical Development, MedImmune
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: D153-P503
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
MeSH Terms: interventions — FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cold-adapted influenza vaccine trivalent (CAIV-T) (Experimental): All subjects were scheduled to receive 2 doses of CAIV-T.The total volume of 0.2 mL was administered intranasally with a spray applicator (approximately 0.1 mL into each nostril).
  Interventions: Biological: CAIV-T

INTERVENTIONS:
Biological: CAIV-T — Each dose of the vaccine was formulated to contain approximately 1 x 10^7 TCID50 of each of three (two subtype A and one subtype B) reassortant 6:2 influenza strains, as described above, for a total of ~3 x 10^7 TCID50 per dose.
  Other Names: FluMist

SUMMARY:
The study was designed to determine the number of doses of CAIV-T required to effectively immunize children and adolescents in the 6 to 17 year age group.

DETAILED DESCRIPTION:
This was a phase II, prospective, open-label, multicenter, outpatient study designed to evaluate the safety, tolerability, and immunogenicity of one or two doses of CAIV-T in children and adolescents between 6 and 17 years of age. Subjects were allocated to one of three study groups according to age at the time of enrollment: study group one consisted of subjects between 6 and 9 years of age, group two of subjects 10 to 12 years of age, and group three of subjects 13 to 17 years of age.

Approximately 450 subjects (ie, 150 subjects per age group) participated in the study and were scheduled to receive two intranasal doses of CAIV-T separated by 35 ± 7 days in an open-label manner.

ELIGIBILITY:
Inclusion Criteria:

* who are at least 6 years and not more than 17 years of age at the time of enrollment;
* who, if female and is post-menarche, has provided a negative pregnancy test; · who are in good health as determined by medical history, physical examination and clinical judgement;
* who have provided written informed consent (as appropriate and according to national guidelines) and whose parent(s) or legal guardian(s) have provided written informed consent after the nature of the study has been explained; 13 who, along with their parent(s) or legal guardian(s), will be available for duration of the study (approximately three months);
* who, together with their parent(s) or legal guardian(s), can be reached by study staff for the post-vaccination contacts [telephone, clinic visit or home visit].

Exclusion Criteria:

* who are perceived to be unavailable or difficult to contact for evaluation or study visits during the study period and whose parent(s) or legal guardian(s) are perceived to be unreliable or difficult to contact for evaluation or study visits during the study period;
* with any serious chronic disease (e.g., with signs of cardiac or renal failure or severe malnutrition), including progressive neurological disease;
* with Down's syndrome or other known cytogenetic disorders;
* with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids;
* who received any blood products, including immunoglobulin, in the period from six months prior to vaccination through to the conclusion of the study;
* for whom there is intent to administer any other investigational vaccine or agent from one month prior to enrollment through to the conclusion of the study;
* have an immunosuppressed or immuno-compromised individual living in the same household;
* who, at any time prior to entry into this study, received a dose of any influenza vaccine (commercial or investigational)
* who, in the two weeks prior to entry into this study, received a dose of any influenza treatment (commercial or investigational)
* with a documented history of hypersensitivity to egg or egg protein or any other component of the study vaccine;
* with a clinically confirmed respiratory illness with wheezing within two weeks prior to enrollment;
* who received aspirin (acetylsalicylic acid) or aspirin-containing products in the two weeks prior to enrollment or for which use is anticipated during the study;
* who were administered any live virus vaccine within one month prior to enrollment or expect receipt of another live virus vaccine within one month of vaccination in this study;
* with any medical conditions that in the opinion of the investigator might interfere with interpretation of the study results; If any of these criteria are met following enrolment, the subject will be excluded from subsequent vaccine dosing.

Note: A pregnant household member is not considered a contraindication to enrollment.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 498 (Actual)
Dates: Start 2000-10; Primary Completion 2001-01 (Actual); Study Completion 2001-01 (Actual)

PRIMARY OUTCOMES:
The number of subjects achieving strain-specific hemagglutination inhibition (HAI) antibody seroconversion post Dose 1 | Day 0, Day 35 post Dose 1
  Immunogenicity was evaluated by comparison of pre and post-vaccination strain-specific titers of serum HAI antibody. Seroconversion was defined as a four-fold or greater rise in serum HAI antibody titer.

SECONDARY OUTCOMES:
The number of subjects achieving strain-specific HAI antibody seroconversion post Dose 1 | Day 0, Day 35 post Dose 2
  Immunogenicity was evaluated by comparison of pre and post-vaccination strain-specific titers of serum HAI antibody. Seroconversion was defined as a four-fold or greater rise in serum HAI antibody titer.
The number of subjects reporting any reactogenicity event post dose | Days 0-10
  Reactogenicity events were predefined adverse events that could have occurred after vaccine administration. They included the following: fever (oral temperature >= 38C), cough, runny nose/nasal congestion, sore throat, irritability, headache, chills, vomiting, decreased activity, decreased appetite, and muscle aches.
The number of subjects reporting any adverse event post dose | Days 0-10
  An adverse event (or adverse experience, AE) was defined as any untoward medical occurrence in a subject who was administered a study product.
The number of subjects reporting serious adverse events post dose | Days 0-42
  An adverse event was considered serious (SAE) if it: resulted in death, regardless of cause; was life-threatening (subject was at risk of death as the event occurred); required inpatient hospitalization or prolonged existing hospitalization; resulted in persistent or significant disability/incapacity; or resulted in a congenital anomaly or birth defect (in the offspring of a vaccine recipient, where applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Raburn Mallory, MD, Study Director — MedImmune LLC
Locations (3):
- Belgium (2):
  - University of Antwerp, Antwerp
  - Dienst Jeugdgezondheidszorg, Leuven
- Oulu University Hospital, Oulu, Finland